CLINICAL TRIAL: NCT01694706
Title: Investigation of the Effect of Food and of Increased Gastric pH on the Relative Bioavailability of a Single Oral Dose of 240 mg Faldaprevir in an Open-label, Randomised, Three-way Cross-over Trial in Healthy Subjects
Brief Title: Investigation of Food Effect and Gastric ph Increase on the Bioavailability of Faldapravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1220.59; 2012-002941-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir; Omeprazole

ARMS (3):
- Reference (Experimental): faldaprevir medium, fasted
  Interventions: Drug: faldaprevir
- Test 1 (Active Comparator): faldaprevir medium, fed
  Interventions: Drug: faldaprevir
- Test 2 (Active Comparator): faldaprevir medium + omeprazole medium
  Interventions: Drug: omeprazole; Drug: faldaprevir

INTERVENTIONS:
Drug: faldaprevir — medium dose of faldaprevir
  Arms: Test 1
Drug: faldaprevir — medium dose of faldaprevir
  Arms: Reference
Drug: omeprazole — medium dose of omeprazole
  Arms: Test 2
Drug: faldaprevir — medium dose of faldaprevir
  Arms: Test 2

SUMMARY:
The primary objective of this trial is to investigate the effect of food and of gastric pH increase on the relative bioavailability of faldaprevir.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.59.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised open label, 3-way cross over study with three sequences. Faldaprevir administrations in each treatment period were separated by washout period of at least 14 days.
Groups:
- Faldaprevir/Faldaprevir+ OMP/Faldaprevir Fed: Faldaprevir: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally following an overnight or at least 10 hours (h) fast prior the drug administration.
  Faldaprevir+ OMP: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast prior the drug administration following multiple dosing of 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir.
  Faldaprevir fed: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally 30 minutes (min) after a standard high-fat, high-caloric meal was served. The meal had to be completely consumed within 25 min or less.
- Faldaprevir Fed/ Faldaprevir/ Faldaprevir+ OMP: Faldaprevir fed: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally 30 minutes (min) after a standard high-fat, high-caloric meal was served. The meal had to be completely consumed within 25 min or less.
  Faldaprevir: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally following an overnight or at least 10 hours (h) fast prior the drug administration (Reference treatment)
  faldaprevir+ OMP: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast prior the drug administration following multiple dosing of 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir.
- Faldaprevir+ OMP/ Faldaprevir Fed/ Faldaprevir: Faldaprevir+ OMP: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast prior the drug administration following multiple dosing of 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir.
  Faldaprevir fed: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally 30 minutes (min) after a standard high-fat, high-caloric meal was served. The meal had to be completely consumed within 25 min or less.
  Faldaprevir: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally following an overnight or at least 10 hours (h) fast prior the drug administration
Period: Overall Study
Arm/Group | Faldaprevir/Faldaprevir+ OMP/Faldaprevir Fed | Faldaprevir Fed/ Faldaprevir/ Faldaprevir+ OMP | Faldaprevir+ OMP/ Faldaprevir Fed/ Faldaprevir
Started | 5 | 5 | 5
Received Faldaprevir | 5 | 5 | 5
Received Faldaprevir +OMP | 5 | 5 | 5
Received Faldaprevir Fed | 4 | 5 | 5
Completed | 4 | 4 | 5
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — other reason not defined above | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) including all subjects who received at least 1 dose of study drug
Groups:
- Entire Study Population: All subjects received all tested treatments in a randomised, open label, 3-way cross over study. The treatments were:
  Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally following an overnight or at least 10 hours (h) fast prior the drug administration (Reference treatment)
  Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally 30 minutes (min) after a standard high-fat, high-caloric meal was served. The meal had to be completely consumed within 25 min or less.
  Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast prior the drug administration following multiple dosing of 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir.
  Drug administrations were separated by a washout period of at least 14 days
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Faldaprevir: Area Under the Curve Over the Time Interval From 0 Extrapolated to Infinity (AUC 0-infinity)
Description: Area under the concentration-time curve of the faldaprevir in plasma over the time interval from 0 extrapolated to infinity
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1.5 hours (h) before drug administration and 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 96h and 120h after drug administration
Population: Pharmacokinetic (PK) set: Included all treated subjects that provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of the pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng*h/mL]
Groups:
- Faldaprevir in Fasting: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally following an overnight or at least 10 hours (h) fast prior the drug administration (Reference treatment)
- Faldaprevir After a High-fat Meal: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was administered orally 30 minutes (min) after a standard high-fat, high-caloric meal was served. The meal had to be completely consumed within 25 min or less
- Faldaprevir and Omeprazole: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast prior the drug administration following multiple dosing of 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir
Arm/Group | Faldaprevir in Fasting | Faldaprevir After a High-fat Meal | Faldaprevir and Omeprazole
Number analyzed (Participants) | 14 | 14 | 14
[ng*h/mL] | 37900 (67.2) | 48200 (41.7) | 36000 (63.4)
Statistical Analysis 1: Comparison: Faldaprevir in Fasting vs Faldaprevir After a High-fat Meal; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.3420, ANOVA; Ratio calculated as Faldaprevir after a high-fat meal divided by Faldaprevir in fasting; Geometric Mean Ratio = 120.35, 90% CI 2-sided [102.09 to 141.88], Standard Deviation 23.2 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Faldaprevir in Fasting vs Faldaprevir and Omeprazole; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.0962, ANOVA; Ratio calculated as Faldaprevir and Omeprazole divided by Faldaprevir in fasting; Geometric Mean Ratio = 94.33, 90% CI 2-sided [76.21 to 116.76], Standard Deviation 30.8 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Faldaprevir: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the faldaprevir in plasma
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Faldaprevir in Fasting | Faldaprevir After a High-fat Meal | Faldaprevir and Omeprazole
Number analyzed (Participants) | 14 | 14 | 14
ng/mL | 2030 (140) | 2600 (57.5) | 1920 (122)
Statistical Analysis 1: Comparison: Faldaprevir in Fasting vs Faldaprevir After a High-fat Meal; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.3993, ANOVA; Ratio calculated as Faldaprevir after a high-fat meal divided by Faldaprevir in fasting; Geometric Mean Ratio = 118.79, 90% CI 2-sided [83.190 to 169.628], Standard Deviation 52.4 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Faldaprevir in Fasting vs Faldaprevir and Omeprazole; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.2204, ANOVA; Ratio calculated as Faldaprevir and Omeprazole divided by Faldaprevir in fasting; Geometric Mean Ratio = 93.55, 90% CI 2-sided [65.783 to 133.030], Standard Deviation 53.0 — Standard deviation is actually the geometric coefficient of variation (gCV)

3. Secondary Outcome: Faldaprevir: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the faldaprevir in plasma over the time interval from 0 to the last quantifiable drug plasma concentration
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Faldaprevir in Fasting | Faldaprevir After a High-fat Meal | Faldaprevir and Omeprazole
Number analyzed (Participants) | 14 | 14 | 14
ng*h/mL | 36300 (70.3) | 46400 (42.6) | 34400 (65.6)
Statistical Analysis 1: Comparison: Faldaprevir in Fasting vs Faldaprevir After a High-fat Meal; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.3765, ANOVA; Ratio calculated as Faldaprevir after a high-fat meal divided by Faldaprevir in fasting; Geometric Mean Ratio = 121.28, 90% CI 2-sided [102.32 to 143.74], Standard Deviation 24.0 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Faldaprevir in Fasting vs Faldaprevir and Omeprazole; Test type: Non-Inferiority or Equivalence — no formal testing, investigation of bioavailability; p = 0.0946, ANOVA; Ratio calculated as Faldaprevir and Omeprazole divided by Faldaprevir in fasting; Geometric Mean Ratio = 94.72, 90% CI 2-sided [76.25 to 117.67], Standard Deviation 31.4 — Standard deviation is actually the geometric coefficient of variation (gCV)

ADVERSE EVENTS:
Time Frame: From first drug administration until the end of trial visit, up until 20 days
Groups:
- Faldaprevir and Omeprazole: Single dose of 240 mg faldaprevir in a form of two soft gelatin capsules was coadministered orally with 40 mg Omeprazole following an overnight or at least 10 hours (h) fast
- Omeprazole: 40 mg omeprazole once daily for 4 days prior the first dose of faldaprevir
Arm/Group | Faldaprevir in Fasting | Faldaprevir After a High-fat Meal | Faldaprevir and Omeprazole | Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 4/14 | 4/14 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir in Fasting (N=15) | Faldaprevir After a High-fat Meal (N=14) | Faldaprevir and Omeprazole (N=14) | Omeprazole (N=15)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes